CLINICAL TRIAL: NCT03289208
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of MCI-186 in Subjects With Mild or Moderate Renal Impairment Compared to Subjects With Normal Renal Function
Brief Title: Pharmacokinetics Study of MCI-186 in Subjects With Mild or Moderate Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MCI-186-J22
Record Dates: First submitted 2017-09-19; First posted 2017-09-20 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Renal Impairment; Healthy
MeSH Terms: conditions — Renal Insufficiency | interventions — Edaravone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mild renal impairment (Experimental)
  Interventions: Drug: MCI-186
- moderated renal impairment (Experimental)
  Interventions: Drug: MCI-186
- normal renal function (Experimental)
  Interventions: Drug: MCI-186

INTERVENTIONS:
Drug: MCI-186 — 30 mg of edaravone will be administered intravenously over 60 minutes.
  Other Names: Edaravone; Radicut

SUMMARY:
To assess the pharmacokinetics of MCI-186 after a single intravenous infusion of 30mg/hour in subjects with mild or moderate renal impairment compared to subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Able to provide written informed consent to participate in this study after reading the ICF
* Subjects is able to understand and willing to cooperate and comply with the Protocol restrictions and requirements
* A body weight of ≥45 kg in males or ≥40 kg in females and a body mass index ranging from 18 to 30 kg/m2

Renal impaired subjects (in addition)

* Subjects with mild renal impairment defined as eGFR 60-89 mL/min/1.73m2 and subjects with moderate renal impairment defined as eGFR 30-59 mL/min/1.73m2
* Chronic and stable renal impairment

Healthy subjects (in addition)

* Subject with normal renal function defined as eGFR≥90 mL/min/1.73m2
* Good health and free from clinically significant illness or disease

Exclusion Criteria:

All subjects

* Presence or history of severe allergy to food, or any medicinal product or relevant excipient that is of clinical significance
* Subjects were previously administered MCI-186
* Positive urine drug screen (if not due to concomitant medication) or alcohol test
* History of alcohol abuse or drug abuse
* Presence of active infection requiring antibiotics
* Positive test for human immunodeficiency virus (HIV) antigen/antibody, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCVAb)

Renal impairment subject (in addition)

* Acute renal failure
* History of renal transplantation
* Aspartate aminotransferase (AST) activity, or an alanine aminotransferase (ALT) activity of at least 3 times the upper limit of normal (ULN) range
* Uncontrolled, or untreated hypertension defined as systolic blood pressure (SBP)>180 mmHg and/or diastolic blood pressure (DBP)>110 mmHg
* Start of any new medication or new any changes to a current dosage

Healthy subject (in addition)

* History or presence of any renal disease
* Uncontrolled, or untreated hypertension defined as systolic blood pressure (SBP)>160 mmHg and/or diastolic blood pressure (DBP)>100 mmHg

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational site, Tokyo, Japan

REFERENCES:
- [Derived] Nakamaru Y, Kakubari M, Yoshida K, Akimoto M, Kondo K. An Open-label, Single-dose Study to Evaluate the Pharmacokinetic Variables of Edaravone in Subjects with Mild, Moderate, or No Renal Impairment. Clin Ther. 2020 Sep;42(9):1699-1714. doi: 10.1016/j.clinthera.2020.06.020. Epub 2020 Aug 28. PMID 32868037

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild Renal Function Group: Mild renal function defined as eGFR 60-89 mL/min/1.73m^2
- Moderate Renal Function Group: Moderate renal function defined as eGFR 30-59 mL/min/1.73m^2
- Normal Renal Function Group: Normal renal function defined as eGFR ≥90 mL/min/1.73m^2
Period: Overall Study
Arm/Group | Mild Renal Function Group | Moderate Renal Function Group | Normal Renal Function Group
Started | 11 | 8 | 11
Completed | 10 | 8 | 11
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Renal Function Group | Moderate Renal Function Group | Normal Renal Function Group | Total
Number analyzed (Participants) | 11 | 8 | 11 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (5.1) | 57.9 (8.4) | 47.3 (4.3) | 45.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 9
  Male | 6 | 6 | 9 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 8 | 11 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Time Frame: pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mild Renal Function Group | Moderate Renal Function Group | Normal Renal Function Group
Number analyzed (Participants) | 6 | 8 | 8
ng/mL | 545.4 (92.59) | 593.2 (115.4) | 475.9 (95.32)

2. Primary Outcome: AUC0-last
Time Frame: pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Mild Renal Function Group | Moderate Renal Function Group | Normal Renal Function Group
Number analyzed (Participants) | 6 | 8 | 8
ng*hr/mL | 758 (148.09) | 808.7 (152.01) | 638.09 (151.98)

3. Primary Outcome: AUC0-∞
Time Frame: pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Mild Renal Function Group | Moderate Renal Function Group | Normal Renal Function Group
Number analyzed (Participants) | 6 | 8 | 8
ng*hr/mL | 770.97 (153.63) | 826.44 (149.44) | 644.85 (153.14)

4. Secondary Outcome: t½
Time Frame: pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Mild Renal Function Group | Moderate Renal Function Group | Normal Renal Function Group
Number analyzed (Participants) | 6 | 8 | 8
hour | 5.38 (6.04) | 7.31 (5.83) | 2.87 (0.38)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Mild Renal Function Group | Moderate Renal Function Group | Normal Renal Function Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 0/8 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mild Renal Function Group (N=11) | Moderate Renal Function Group (N=8) | Normal Renal Function Group (N=11)
Bronchitis (Infections and infestations) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Vomitting (Gastrointestinal disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT03289208/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03289208/SAP_001.pdf